CLINICAL TRIAL: NCT01000597
Title: An Open-label, Randomised, Two-way Crossover Study, to Evaluate and Compare the Pharmacokinetics of Fluticasone Furoate, Administered From a Novel Dry Powder Device (Repeat Dose) and Intravenously (Single Dose), in Healthy Caucasian, Japanese, Korean and Chinese Subjects
Brief Title: Study to Look at and Compare How Inhaled and Intravenous Fluticasone Furoate is Processed by the Body in Healthy Caucasian, Japanese, Korean and Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 113477
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: pharmacokinetics; serum cortisol; pharmacodynamics; fluticasone furoate; healthy Caucasian, Japanese, Korean and Chinese subjects
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Y (Other): Seven inhaled doses of 200mcg FF given once daily in the morning (Part A; Days 1-7) followed by seven inhaled doses of 800mcg FF given once daily in the morning (Part B; Day 1 and Days 3-8, i.e. no dose on Day 2).
  Interventions: Drug: fluticasone furoate
- Treatment Z (Other): A single intravenous dose of 250mcg FF given over 20 minutes (Day 1).
  Interventions: Drug: fluticasone furoate

INTERVENTIONS:
Drug: fluticasone furoate — Seven inhaled doses of 200mcg FF given once daily in the morning (Part A; Days 1-7) followed by seven inhaled doses of 800mcg FF given once daily in the morning (Part B; Day 1 and Days 3-8, i.e. no dose on Day 2).
  A single intravenous dose of 250mcg FF given over 20 minutes (Day 1).

SUMMARY:
Previous studies have shown potentially higher exposure to fluticasone furoate in Japanese subjects compared with Caucasian subjects. The reasons for these potential differences are unclear. Therefore this study is being done to look at and compare how fluticasone furoate is processed by the body in healthy Caucasian, Japanese, Korean and Chinese subjects after inhaled and intravenous administration. The data obtained will be used to help in the clinical development of the drug in Japanese and other East Asian populations.

DETAILED DESCRIPTION:
Corticosteroids are a highly effective anti-inflammatory therapy in allergic conditions such as asthma and rhinitis. Fluticasone Furoate (FF) is a novel corticosteroid with potent glucocorticoid activity similar to fluticasone propionate and mometasone furoate. Phase II studies have shown FF to be an effective once daily inhaled steroid for asthma and it is being developed as a potential steroid component in a once daily combination with GW642444M, for once-daily administration for the maintenance treatment of asthma and COPD. FF is approved worldwide (including the US, EU and Japan) as an intranasal steroid for the treatment of allergic rhinitis (VERAMYST™ /AVAMYS™ /ALLERMIST™). Previous inter-study comparisons have indicated potentially higher systemic exposure to FF in Japanese subjects compared with treatment groups that recruited predominantly Caucasian subjects. The reasons for these potential differences are unclear. This study is being performed to evaluate and directly compare the PK and systemic PD effects of FF in healthy Caucasian, Japanese, Korean and Chinese subjects when delivered from the novel dry powder inhaler and intravenously. The data obtained will be used to facilitate clinical development of the FF/GW642444 combination in Japanese and other East Asian populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between 20 and 64 years of age inclusive
* Caucasian, Japanese, Korean or Chinese
* Body mass index (BMI) for Caucasians within the range 18.5-29.0 kg/m2 (inclusive). For East Asians BMI within the range 18.5-24.9 kg/m2 (inclusive) and height 1.55m-1.85m (inclusive)
* Non-smokers
* AST, ALT, alkaline phosphatase and bilirubin </=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* No significant abnormality on 12-lead ECG at screening
* No significant abnormality on the Holter ECG at screening
* FEV1 >/= 85% predicted at screening
* Capable of giving written informed consent
* Subjects who are able to use the inhalation device satisfactorily

Exclusion Criteria:

* As a result of screening medical exam, the principal investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age.
* Any history of breathing problems in adult life
* Pregnant or lactating females
* Subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of milk protein allergy.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Subject has taken oral corticosteroids less than 8 weeks before the screening visit.
* Subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* History of alcohol/drug abuse or dependence within 12 months of the study
* Subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Positive for HIV antibodies.
* Positive pre-study urine drug screen or when randomly tested during the study.
* Positive carbon monoxide or alcohol breath test at screening or on admission to the Unit.
* Positive urine cotinine test at screening.
* Consumption of seville oranges, pomelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09-17 (Actual); Primary Completion 2009-12-23 (Actual); Study Completion 2009-12-23 (Actual)

PRIMARY OUTCOMES:
FF Pharmacokinetic parameters: AUC, Cmax, t1/2, tmax for inhaled and intravenous treatments. Volume of distribution (V) and plasma clearance (CL) for intravenous FF | up to 72hr PK sampling periods profiles on 4 separate occasions over a total period of approximately 4-5 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters MRT for both inhaled and intravenous treatments; MAT, AUC(0-t) for 200mcg dose,observed accumulation (Ro) and absolute bioavailability for inhaled treatment | up to 72hr PK sampling periods profiles on 4 separate occasions over a total period of approximately 4-5 weeks
Pharmacodynamics; serum cortisol for 200mcg inhaled FF treatment only: 24 hour weighted mean (on Day -1 and Day 7) | Two 24 hour sampling periods approximately 1 week apart
• Ratio of twenty-four hour urine cortisol to 6-beta-hydroxy-cortisol (on Day -1 of first treatment period only). Plasma 4-beta-hydroxy-cholesterol (single sample, on Day -1 of first treatment period only). Measure of baseline CYP3A4 activity | One collection period of up to 24 hours
• Vital signs, 12-lead ECG, Clinical laboratory tests, forced expiratory volume in 1 second (FEV1) (at screening), peak expiratory flow rate (PEFR), AEs. | Throughout study; approx 10 weeks
Quantity of the total emitted dose (TED), ex-throat dose (ETD) and mass less than 2 micrometer of inhaled FF for each subject, assessed by pharyngometry, inhalation profile, breath hold and lung volume measurements | Throughout study from screening to end of treatment periods; approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113477 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113477?search=study&search_terms=113477#rs
- Available data/document: Statistical Analysis Plan: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113477 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register